CLINICAL TRIAL: NCT06079177
Title: B-lines Score Derived From Lung Ultrasonography as a Noninvasive Indicator for the Systemic Volumetric Load During TURP. A Prospective Observational Study.
Brief Title: B-lines Score as Indicator for the Systemic Volumetric Load During TURP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dalia Saad Abd-El Kader, assistant professor, Kasr El Aini Hospital
Other Study IDs: MD-295/2022
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Transurethral Resection of Prostate
Keywords: Lung Ultrasonography score (LUS); extravascular lung water (EVLW); Transurethral resection of the prostate (TURP)
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients with age ≥ 60 years undergoing TURP surgery: All patients will receive spinal anesthesia Under complete aseptic technique at level of L 4-L5 or L3-L4 using 12.5-15 mg of 0.5 % hyperbaric bupivacaine and 25 ug fentanyl.
  Lung ultrasound score:
  A curvilinear (5-2 MHz) probe will be used. The sliding multiple B-lines will be evaluated in eight antero-lateral lung examination zones.
  Inferior vena cava (IVC) measurement using ultrasound:
  A curvilinear (5-2 MHz) probe with B-mode scan will be used. Caval-Aorta index will be calculated by taking the ratio of the two respective diameters measured.
  Other vital parameter as ,heart rate (HR), Mean arterial pressure (MAP), oxygen saturation (SpO2), arterial blood gases (ABG), serum Na and K levels will be measured and recorded at same time as the following:
  (T0) ,(T1) ,(T2),(T3) ,(T30, T60, T90) intraoperative ,(T PACU),(T critical)
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — LUS using B-lines Caval-Aorta index using ultrasound

SUMMARY:
Lung Ultrasonography score (LUS) using B-lines is a noninvasive, reliable and promising method for determining the extravascular lung water (EVLW). This was previously evaluated by trans-pulmonary thermodilution technique.

The transurethral resection of the prostate syndrome (TURP-S) is a potentially life-threatening complication of the TURP surgery and timely diagnosis of TURP-S is crucial for rapid detection and optimized treatment.

This observational study is designed to investigate the use of LUS using B-lines as a bed-side, simple, and non-invasive indicator for predication of the presence of systemic volume overload in patients undergoing endoscopic TURP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years.
* American Society of Anesthesiologists Classification (ASA ) I, II, and III.
* Full conscious patients.

Exclusion Criteria:

* Patient refusal.
* Who known allergic or hypersensitivity to any drug used in the study (local anesthesia).
* Coagulopathy (history of bleeding disorders), or patients on anticoagulant drugs, with (platelets <50,000 International Normalised Ratio( INR)>1.5).
* Patients have renal dysfunction patients with creatinine ≥ 2.
* Patients have uncontrolled cardiac diseases (IHD, (congestive heart failure (CHF), pulmonary hypertension and valvular diseases).
* Abdominal ascites.
* Patients with local infection at the site of local anesthetic injection.
* Failed spinal anesthesia.
* Timing not exceed 90 min.
* Any patient with lung ultrasound examination at T 0 ≥ 3 B-lines will be excluded from the study.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male patients with age ≥ 60 years undergoing TURP surgery
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Predictive ability of the LUS using B-lines for the presence of systemic volume overload in patients undergoing endoscopic TURP | From the preoperative period (T0) to 60 Minutes postoperative (T PACU)
  using ultrasound

SECONDARY OUTCOMES:
Predictive ability of the Caval-Aorta index as predictors of systemic volume overload in patients undergoing endoscopic TURP. | From the preoperative period (T0) to 60 Minutes postoperative (T PACU)
  using ultrasound
Correlation between the absolute value of LUS, Caval-Aorta index . | From the preoperative period (T0) to 60 Minutes postoperative (T PACU)
  using ultrasound
Correlation between the relative changes of the LUS and Caval-Aorta index | From the preoperative period (T0) to 60 Minutes postoperative (T PACU)
  using ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Saad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demirel I, Ozer AB, Bayar MK, Erhan OL. TURP syndrome and severe hyponatremia under general anaesthesia. BMJ Case Rep. 2012 Nov 19;2012:bcr-2012-006899. doi: 10.1136/bcr-2012-006899. PMID 23166168
- [Background] Rassweiler J, Teber D, Kuntz R, Hofmann R. Complications of transurethral resection of the prostate (TURP)--incidence, management, and prevention. Eur Urol. 2006 Nov;50(5):969-79; discussion 980. doi: 10.1016/j.eururo.2005.12.042. Epub 2006 Jan 30. PMID 16469429
- [Background] Nakahira J, Sawai T, Fujiwara A, Minami T. Transurethral resection syndrome in elderly patients: a retrospective observational study. BMC Anesthesiol. 2014 Apr 23;14:30. doi: 10.1186/1471-2253-14-30. eCollection 2014. PMID 24782656
- [Background] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866
- [Background] El-Baradey GF, El-Shmaa NS. Does caval aorta index correlate with central venous pressure in intravascular volume assessment in patients undergoing endoscopic transuretheral resection of prostate? Saudi J Anaesth. 2016 Apr-Jun;10(2):174-8. doi: 10.4103/1658-354X.168062. PMID 27051368
- [Background] Anile A, Russo J, Castiglione G, Volpicelli G. A simplified lung ultrasound approach to detect increased extravascular lung water in critically ill patients. Crit Ultrasound J. 2017 Dec;9(1):13. doi: 10.1186/s13089-017-0068-x. Epub 2017 Jun 13. PMID 28612302
- [Background] Volpicelli G, Skurzak S, Boero E, Carpinteri G, Tengattini M, Stefanone V, Luberto L, Anile A, Cerutti E, Radeschi G, Frascisco MF. Lung ultrasound predicts well extravascular lung water but is of limited usefulness in the prediction of wedge pressure. Anesthesiology. 2014 Aug;121(2):320-7. doi: 10.1097/ALN.0000000000000300. PMID 24821071
- [Background] Salama ER, Elkashlan M. Pre-operative ultrasonographic evaluation of inferior vena cava collapsibility index and caval aorta index as new predictors for hypotension after induction of spinal anaesthesia: A prospective observational study. Eur J Anaesthesiol. 2019 Apr;36(4):297-302. doi: 10.1097/EJA.0000000000000956. PMID 30664523